CLINICAL TRIAL: NCT06419816
Title: A Primary Care-Based, Prospective, Multicenter, Cluster-Randomized, Pragmatic Clinical Trials to Determine the Effect of Linking Data With Investigators When Using the Electronic Health Record-Linked Smartphone Application, 'Well Check', on Clinical Outcomes in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Linking Data Using Smartphone Application, 'Well Check', on Clinical Outcomes in Patients With Type 2 Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_ODNENV_DB_01
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes: mobile application "WellCheck" use
  Interventions: Other: Physician-managed "WellCheck" use; Other: self-managed "WellCheck" use

INTERVENTIONS:
Other: Physician-managed "WellCheck" use — Physician-managed "WellCheck" use
Other: self-managed "WellCheck" use — self-managed "WellCheck" use

SUMMARY:
This clinical study aims to evaluate the effects of using the "WellCheck" mobile application on blood glucose, blood pressure, and weight among Type 2 diabetes patients in real primary care settings. It is a prospective, multi-center, cluster-randomized, pragmatic clinical trial. Patients who can use the digital healthcare mobile application without difficulty are recruited based on the clinical judgment of the attending physician.

DETAILED DESCRIPTION:
The study employs a 1:1 cluster-randomized allocation to differentiate between intervention (physician-managed "WellCheck" use) and control groups (self-managed "WellCheck" use) within primary care facilities where intervention and control groups are treated separately. Data collection includes demographic information, physical measurements, vital signs, laboratory tests, and safety evaluations for up to 24 weeks following the initiation of "WellCheck" use. While data collection aligns with routine clinical practice, additional follow-up visits are scheduled at 6, 12, 18, and 24 weeks post-baseline for efficacy and safety assessments. Researchers will collect necessary data based on routine clinical records and "WellCheck" data.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years and older.
2. Patients with Type 2 diabetes who are scheduled to receive initial treatment with Enavogliflozin or Enavogliflozin Extended-Release Tablets based on the attending physician's medical judgment, within the following insurance coverage ranges:

   * Enavogliflozin monotherapy
   * Combination therapy of Enavogliflozin with two agents (metformin)
   * Combination therapy of Enavogliflozin with three agents (metformin + DPP-4 inhibitor)
3. Individuals who have received detailed explanation and have understood the nature of the observational study and the investigational drug, and have provided written consent to participate voluntarily in the observational study and to comply with subject precautions during the study period.

Exclusion Criteria:

1. Individuals with diabetes other than Type 2 diabetes (Type 1 diabetes, diabetic ketoacidosis, gestational diabetes, etc.).
2. Individuals who are contraindicated for Enavogliflozin or Enavogliflozin Extended-Release Tablets based on the approved indications:

   * Patients with a history of hypersensitivity reactions to the components of Enavogliflozin or Enavogliflozin Extended-Release Tablets
   * Patients with an eGFR (estimated Glomerular Filtration Rate) less than 30 mL/min/1.73m2, end-stage renal disease, or undergoing dialysis
   * Patients with moderate to severe hepatic impairment (AST or ALT > 3 times the upper limit of normal, Total Bilirubin > 2 times the upper limit of normal, hepatitis or hepatic failure)
   * Patients classified as NYHA (New York Heart Association) class III or IV
3. Patients initiating treatment with Enavogliflozin or Enavogliflozin Extended-Release Tablets at enrollment with an eGFR of less than 60ml/min/1.73m2.
4. Patients with unstable weight due to treatment with obesity drugs or weight loss medications within 3 months prior to enrollment or other treatments (surgery, dietary therapy, etc.).
5. Pregnant and lactating women.
6. Individuals currently participating in another clinical trial and receiving investigational drugs or investigational medical devices.
7. Other individuals deemed unsuitable for participation in the observational study based on the investigator's (attending physician's) judgment.

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: According to the calculation using G*Power 3.1.9.7, the required sample size for conducting this study is determined to be 11,698 individuals. Considering an approximate dropout rate of 30%, recruitment of around 15,000 participants is planned.
Sampling Method: Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
change in glycated hemoglobin (HbA1c) levels | 24 weeks
  change in glycated hemoglobin (HbA1c) levels at 24 weeks from baseline

SECONDARY OUTCOMES:
change in glycated hemoglobin (HbA1c) levels | 6 weeks
  change in glycated hemoglobin (HbA1c) levels at 6 weeks post-baseline
change in glycated hemoglobin (HbA1c) levels | 12 weeks
  change in glycated hemoglobin (HbA1c) levels at 12 weeks post-baseline
change in glycated hemoglobin (HbA1c) levels | 18 weeks
  change in glycated hemoglobin (HbA1c) levels at 18 weeks post-baseline
the change in fasting plasma glucose (FPG) | 6 weeks
  the change in fasting plasma glucose (FPG) at 6 weeks post-baseline
the change in fasting plasma glucose (FPG) | 12 weeks
  the change in fasting plasma glucose (FPG) at 12 weeks post-baseline
the change in fasting plasma glucose (FPG) | 18 weeks
  the change in fasting plasma glucose (FPG) at 18 weeks post-baseline
the proportion of participants achieving HbA1c less than 7% or 6.5% | 6 weeks
  the proportion of participants achieving HbA1c less than 7% or 6.5% at 6 weeks post-baseline
the proportion of participants achieving HbA1c less than 7% or 6.5% | 12 weeks
  the proportion of participants achieving HbA1c less than 7% or 6.5% at 12 weeks post-baseline
the proportion of participants achieving HbA1c less than 7% or 6.5% | 18 weeks
  the proportion of participants achieving HbA1c less than 7% or 6.5% at 18 weeks post-baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sang H, Kim S, Hwang J, Woo S, Hwang Y, Kim J, Lee S, Yon DK, Rhee SY. Impact of the WellCheck smartphone app linked to electronic health records on clinical outcomes in patients with type 2 diabetes: Study protocol for primary care-based, prospective, multicenter, cluster-randomized, pragmatic clinical trials. PLoS One. 2025 Aug 7;20(8):e0329003. doi: 10.1371/journal.pone.0329003. eCollection 2025. PMID 40773465